CLINICAL TRIAL: NCT05299606
Title: A Prospective Multicenter Study of Transbronchial Microwave Ablation Using Robotic-Assisted Bronchoscopy in Subjects With Oligometastatic Tumors in the Lung
Brief Title: POWER Study (Prospective Transbronchial Microwave + Robotic-Assisted Bronchoscopy)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in Sponsor strategy
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU_2020_03
Record Dates: First submitted 2022-03-03; First posted 2022-03-29 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transbronchial Microwave Ablation (Experimental): Transbronchial microwave ablation will be performed using the NEUWAVE FLEX Microwave Ablation System and Accessories on oligometastatic tumors in the peripheral lung, guided by the Auris MONARCH Platform for visualization and access while using cone beam CT (computed tomography) to confirm probe tip placement and final ablation zone.
  Interventions: Device: Transbronchial Microwave Ablation

INTERVENTIONS:
Device: Transbronchial Microwave Ablation — Transbronchial microwave ablation will be performed using the NEUWAVE FLEX Microwave Ablation System and Accessories on oligometastatic tumors in the peripheral lung, guided by the Auris MONARCH Platform for visualization and access while using cone beam CT (computed tomography) to confirm probe tip placement and final ablation zone.

SUMMARY:
This is a prospective, multicenter, single-arm study on transbronchial microwave ablation using the NEUWAVE FLEX Microwave Ablation System and Accessories on oligometastatic tumors in the peripheral lung, guided by the Auris MONARCH Platform for visualization and access while using cone beam CT (computed tomography) to confirm probe tip placement and final ablation zone. The primary endpoint is Technique Efficacy, assessed 30-days post-ablation via CT imaging.

ELIGIBILITY:
INCLUSION CRITERIA:

* Signed informed consent.
* Subjects greater or equal to 22 years old.
* Performance status 0-2 (Eastern Cooperative Oncology Group classification (ECOG).
* Willing to fulfill all follow-up visit requirements.
* Subjects with at least one oligometastatic lung tumor where the primary tumor is controlled (in the opinion of the investigator or treating oncologist).
* Oligometastatic lung tumor(s) planned to be ablated in the outer two-thirds of the lung and not closer than 1cm to the pleura.

EXCLUSION CRITERIA:

* Pregnant or breastfeeding.
* Subjects with thoracic implantable devices, including pacemakers or other electronic implants.
* Chronic, continuous ventilator support, which uses bi-level positive airway pressure (PAP) to improve lung function for severe conditions. (However, intermittent PAP, for non-pulmonary conditions, such as sleep apnea, is permitted).
* Prior pneumonectomy.
* Severe bronchiectasis (with FEV1 <30%) or disease deemed to be too severe in the opinion of the investigator.
* Platelet count ≤ 50,000/mm3.
* Subjects with uncorrectable coagulopathy at time of screening.
* Subjects medically unable to stop anti-platelet agents (e.g., aspirin, clopidogrel, prasugrel, ticagrelor) at least 5 days prior to the procedure through 48-72 hours after the procedure.
* Subjects medically unable to stop warfarin at least 3-5 days prior to the ablation procedure, or until INR < 1.5, through 48-72 hours after the procedure. On the day of the procedure, subjects with an INR > 1.5 cannot have the procedure completed that day but may be rescheduled or postponed.
* Subjects medically unable to stop anticoagulants (e.g., rivaroxaban, apixaban, dabigatran, endoxaban) at least 3 days prior to the ablation procedure through 48-72 hours after the procedure.
* Expected survival less than 6 months in the opinion of the investigator and/or treating oncologist.
* Subjects with known or suspected brain metastases.
* Subject has had any radiation (i.e., SBRT or EBRT) to the intended ablation zone.
* Endobronchial tumors proximal to and including the segmental airways.
* Lung ablation, surgical resection therapy, radiotherapy, or any other treating procedure within 30 days prior to the planned study ablation procedure or those who plan to receive a lung ablation, surgical resection, or radiation therapy on the ablated lung side before completing the primary endpoint assessment (30 days post-ablation).
* Systemic therapy (e.g., chemotherapy, targeted drug therapy, or immunotherapy) within 14 days prior to the planned study ablation procedure or those who plan to receive systemic therapy before completing the primary endpoint assessment (30 days post-ablation).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - Stanford University School of Medicine, Stanford, California
  - UCONN Health, Farmington, Connecticut
  - Minnesota Lung Center, Minneapolis, Minnesota
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson, Houston, Texas
- Canada (2):
  - University of Toronto, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Transbronchial Microwave Ablation: Each participant underwent transbronchial microwave ablation to the target oligometastatic tumor(s) in the peripheral lung. The treating physician used the NEUWAVE FLEX Microwave Ablation System and Accessories, guided by the Auris MONARCH Platform for visualization and access while using cone beam CT (computed tomography) to confirm probe tip placement and final ablation zone. The treating physician determined the ablation time and power used on a case-by-case basis.
Period: Overall Study
Arm/Group | Transbronchial Microwave Ablation
Started | 12
Completed | 11
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: 12 patients were enrolled and treated
Arm/Group | Transbronchial Microwave Ablation
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of patient at the time they signed the Informed Consent Form.
  Years | 53.5 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 1
  Unknown or Not Reported | 1
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 2
  Former Smoker | 7
  Non-Smoker | 3
Primary Cancer Diagnosis [Count of Participants; unit: Participants]
  Colorectal | 8
  Renal | 2
  Sarcoma | 2
Stage at Time of Primary Cancer Diagnosis [Count of Participants; unit: Participants] — Primary cancer (colorectal, renal, or sarcoma) diagnosis stage. A higher stage indicates more advanced cancer. Stage I: Cancer is a small tumor (<4 cm-renal, <5 cm-sarcoma, in inner bowel layers-colorectal) that has not spread to lymph nodes or distant organs.
  Stage II: Cancer is a larger tumor (>4-10 cm-renal, 5-10 cm-sarcoma, in bowel wall outer layers-colorectal) that has not spread to lymph nodes or distant organs.
  Stage III: Cancer may have spread to nearby lymph nodes, but has not spread to distant organs.
  Stage IV: Cancer has spread to distant organs (metastatic or advanced disease).
  Participants
    Stage I | 3
    Stage II | 2
    Stage III | 6
    Stage IV | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Whose Ablation Resulted in Technique Efficacy
Description: Technique Efficacy is defined as ablation of the target tumor(s) with the ablation zone completely overlapping or encompassing the entire target tumor(s) as assessed using CT imaging 30 days (- 7 to +14 days) after the ablation procedure.
Time Frame: 30 days post-ablation
Population: Patients analyzed at 30 days post-ablation. 11 patients were analyzed as 1 patient passed away before the 30 day post-ablation visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Transbronchial Microwave Ablation
Number analyzed (Participants) | 11
Participants | 11

2. Secondary Outcome: Number of Patients Whose Ablation Resulted in Technical Success
Description: Technical Success is defined as ablation of the target lesion(s) according to the protocol and covered completely, with an adequate margin (that is, the ablation zone completely overlaps or encompasses the target lesion plus an ablative margin), as assessed by the performing physician using CBCT imaging, immediately following the procedure.
Time Frame: Immediately post-ablation (Day 0)
Population: All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Transbronchial Microwave Ablation
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: Number of Patients Who Experienced Local Tumor Progression
Description: Local Tumor Progression, or recurrence of the originally ablated tumor(s) within or abutting the ablation zone, using the 30 day post-ablation imaging as baseline, was analyzed at 3 months, 6 months and 1 year post-ablation via CT imaging
Time Frame: Assessed at 3 months, 6 months and 1 year post-ablation
Population: Patients analyzed 30 days post-ablation through the 1 year follow up period. 11 patients were analyzed as 1 patient passed away before the 30 day post-ablation visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Transbronchial Microwave Ablation
Number analyzed (Participants) | 11
Participants | 11

4. Secondary Outcome: Number of Patients Who Experienced Disease Progression
Description: Disease Progression includes local tumor progression (that is, recurrence of the target ablated tumor within or abutting the ablation zone) and regional tumor progression (that is, new or progression of non-ablated pre-existing tumors within the lung but outside the ablation zone) and distant tumor progression. Results for each category (local, regional, and distant tumor progression) are specified, as well as Overall Disease Progression. Disease Progression was analyzed at 3 months, 6 months and 1 year post-ablation via CT imaging as per treating physician assessment
Time Frame: Assessed at 3 months, 6 months and 1 year post-ablation
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transbronchial Microwave Ablation
Number analyzed (Participants) | 11
Participants
  Overall Disease Progression | 3
  Local Tumor Progression | 0
  Regional Tumor Progression | 3
  Distant Tumor Progression | 2

5. Secondary Outcome: Number of Patients Who Required Repeat Ablation of Target Lesion
Description: Number of patients that experienced a recurrence of the successfully ablated target lesion, as assessed at Day 30 post-ablation, and underwent a repeat ablation of the target Lesion
Time Frame: Assessed at 3 months, 6 months and 1 year post-ablation
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transbronchial Microwave Ablation
Number analyzed (Participants) | 11
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year following the initial ablation procedure.
Description: Participants were evaluated for AEs and SAEs at every study visit from the time of consent through the end-of-study (1 year following the initial ablation procedure).
Arm/Group | Transbronchial Microwave Ablation
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transbronchial Microwave Ablation (N=12)
Post-ablation syndrome (Injury, poisoning and procedural complications) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transbronchial Microwave Ablation (N=12)
Post-ablation syndrome (Injury, poisoning and procedural complications) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (Gastrointestinal disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT05299606/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT05299606/SAP_001.pdf